CLINICAL TRIAL: NCT02706899
Title: A Phase 1/2 Study of Vadastuximab Talirine (SGN-CD33A) in Combination With Azacitidine in Patients With Previously Untreated International Prognostic Scoring System (IPSS) Intermediate-2 or High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Study of Vadastuximab Talirine (SGN-CD33A; 33A) in Combination With Azacitidine in Patients With Previously Untreated Higher Risk MDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGN33A-004
Record Dates: First submitted 2016-02-19; First posted 2016-03-11 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Myelodysplastic Syndrome
Keywords: Antibody-Drug Conjugate CD33 Antigen
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — vadastuximab talirine; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 33A + azacitidine (Experimental): Vadastuximab talirine plus azacitidine
  Interventions: Drug: vadastuximab talirine; Drug: Azacitidine
- Placebo + azacitidine (Active Comparator): placebo plus azacitidine
  Interventions: Drug: Azacitidine; Drug: Placebo (for 33A)

INTERVENTIONS:
Drug: vadastuximab talirine — Intravenous (IV) push every 4 weeks
  Other Names: 33A; SGN-CD33A
  Arms: 33A + azacitidine
Drug: Azacitidine — 75 mg/m^2 given intravenously or subcutaneously for 7 days every 4 weeks
Drug: Placebo (for 33A) — Placebo supplied in single-use vials matching 33A, IV push every 4 weeks
  Arms: Placebo + azacitidine

SUMMARY:
This is a phase 1/2 study to evaluate the combination of vadastuximab talirine (SGN-CD33A; 33A) and azacitidine in subjects with previously untreated International Prognostic Scoring System (IPSS) Intermediate-2 or high risk myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
In the phase 1 portion of the study, escalating doses of 33A will be evaluated in combination with azacitidine, and a dose of 33A will be selected to proceed to phase 2. The phase 2 portion of the study is randomized, double-blind and placebo-controlled; it is designed to compare the overall response rate (ORR) between 2 study arms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cytologically/histologically confirmed MDS according to the World Health Organization (WHO) 2008 classification.
* Previously untreated for Myelodysplastic Syndrome (MDS)
* Age ≥18 years of age.
* Eligible for therapy with azacitidine.
* Life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Adequate baseline laboratory parameters.

Exclusion Criteria:

* Received prior treatment for MDS with lenalidomide or hypomethylating agents (HMAs).
* History of one of the following myeloproliferative neoplasms: essential thrombocythemia, polycythemia vera, and primary myelofibrosis.
* Second malignancy currently requiring active therapy (except for hormonal/anti-hormonal treatment, eg, prostate or breast cancer).
* Candidates for allogeneic stem cell transplant at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02; Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Garfin, Study Chair — Seagen Inc.
Locations (34):
- United States (34):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Southern California, Los Angeles, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Colorado Hospital, Denver, Colorado
  - Cancer Specialisits of North Florida, Fleming Island, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Georgia Regents University Hospital, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Medical Center (UMMC), Minneapolis, Minnesota
  - Bozeman Deaconess Health Group, Bozeman, Montana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Weill Cornell, Brooklyn, New York
  - Westchester Medical Center, Hawthorne, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Case Western Reserve University (CWRU) - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence Portland Research Center, Portland, Oregon
  - Oregon Health & Science, Portland, Oregon
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington
  - Froedtert & Medical College of Wisconson Clinical Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- 33A (5 mcg/kg) + Azacitidine: Vadastuximab talirine (33A) plus azacitidine
  Vadastuximab talirine (5mcg/kg) given via intravenous (IV) push every 4 weeks
  Azacitidine (75 mg/m^2) given intravenously or subcutaneously x 7 days every 4 weeks
- 33A (10 mcg/kg) + Azacitidine: Vadastuximab talirine (33A) plus azacitidine
  Vadastuximab talirine (10mcg/kg) given via intravenous (IV) push every 4 weeks
  Azacitidine (75 mg/m^2) given intravenously or subcutaneously x 7 days every 4 weeks
Period: Overall Study
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Started | 13 | 6
Completed | 0 | 0
Not Completed | 13 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 8 | 0
Not completed — Study Termination by Sponsor | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Continuous [Median (Full Range); unit: years] | 72 [46 to 83] | 66 [57 to 81] | 72 [46 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 10 | 5 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed less than 50% of the time; 3= In bed more than 50% of the time; 4=100% bedridden; 5=Dead
  Participants
    Grade 0: Normal activity | 6 | 2 | 8
    Grade 1: Symptoms but ambulatory | 6 | 4 | 10
    Grade 2: In bed less than 50% of the time | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Outcome Measure: Recommended Dose of Vadastuximab Talirine for the Phase 2 Portion of the Study
Description: A recommended dose of vadastuximab talirine was not identified in Phase 1 due to study termination. Number of dose delays and reductions are reported in lieu of a dose recommendation.
Time Frame: Up to 1 year
Measure: Number; unit: Number of doses
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Number analyzed (Participants) | 13 | 6
Number of doses
  Vadastuximab talirine doses delayed | 2 | 0
  Vadastuximab talirine dosed reduced | 4 | 1
  Azacitidine doses delayed | 3 | 3
  Azacitidine doses reduced | 2 | 2
  Azacitidine unplanned dose adjustments | 3 | 0

2. Primary Outcome: Phase 2 Outcome Measure: Overall Response Rate for the Phase 2 Portion of the Study
Time Frame: N/A - End point not assessed
Population: No patients were assessed for this outcomes as the study did not progress to Phase 2.
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Safety of the Combination of Vadastuximab Talirine and Azacitidine Measured by the Number of Participants With Adverse Events and Laboratory Abnormalities
Description: As defined by the number of participants with adverse events and laboratory abnormalities. Participants are included only once per row, even if the participant experienced multiple events applicable to the category.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Number analyzed (Participants) | 13 | 6
Participants
  Treatment-emergent adverse event (TEAE) | 13 | 6
  Vadatuximab talirine-related TEAE | 9 | 6
  Azacitidine-related TEAE | 13 | 6
  Serious TEAE | 9 | 4
  Vadatuximab talirine-related serious TEAE | 4 | 4
  Azacitidine-related serious TEAE | 5 | 4
  TEAE of Grades 3-5 | 12 | 6
  Vadatuximab talirine-related TEAE of Grades 3-5 | 9 | 6
  Azacitidine-related TEAE of Grades 3-5 | 10 | 6
  TEAE with outcome of death | 2 | 0
  Dose-limiting toxicity | 2 | 0

4. Secondary Outcome: Complete Response Rate (CR)
Description: Study did not progress to Phase 2. A comparison between the 2 arms (Phase 2) of the CR rate, as defined by the 2006 IWG criteria for MDS.
Time Frame: N/A - End point not assessed
Population: No patients were assessed for this outcomes as the study did not progress to Phase 2.
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Hematologic Improvement (HI) Rate
Description: Study did not progress to Phase 2. A comparison between the 2 arms (Phase 2) of the HI rate, as defined by the 2006 IWG criteria for MDS.
Time Frame: N/A - End point not assessed
Population: No patients were assessed for this outcomes as the study did not progress to Phase 2.
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response (DOR) Rate
Description: Study did not progress to Phase 2. A comparison between the 2 arms (Phase 2) of the time from first observation of response (CR, PR, or Marrow CR) to disease progression/relapse or death from any cause, whichever occurs first.
Time Frame: N/A - End point not assessed
Population: No patients were assessed for this outcomes as the study did not progress to Phase 2.
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Progression Free Survival (PFS)
Description: Study did not progress to Phase 2. A comparison between the 2 arms (Phase 2) of the time from first dose of study medication to first documentation of disease progression/relapse, or to death due to any cause, whichever occurs first.
Time Frame: N/A - End point not assessed
Population: No patients were assessed for this outcomes as the study did not progress to Phase 2.
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Rate of Transformation to Acute Myeloid Leukemia (AML)
Description: Study did not progress to Phase 2. A comparison between the 2 arms (Phase 2) of the rate of transformation to AML after initiation of study therapy.
Time Frame: N/A - End point not assessed
Population: No patients were assessed for this outcomes as the study did not progress to Phase 2.
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Overall Survival (OS)
Description: Study did not progress to Phase 2. A comparison between the 2 arms (Phase 2) of the time from first dose of study medication to death due to any cause.
Time Frame: N/A - End point not assessed
Population: No patients were assessed for this outcomes as the study did not progress to Phase 2.
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Treatment-emergent adverse events: a newly occurring or worsening adverse event after the first dose of study drug.
Arm/Group | 33A (5 mcg/kg) + Azacitidine | 33A (10 mcg/kg) + Azacitidine
All-Cause Mortality (participants affected / at risk) | 8/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 9/13 | 4/6
Other Adverse Events (participants affected / at risk) | 13/13 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 33A (5 mcg/kg) + Azacitidine (N=13) | 33A (10 mcg/kg) + Azacitidine (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 33A (5 mcg/kg) + Azacitidine (N=13) | 33A (10 mcg/kg) + Azacitidine (N=6)
Nausea (Gastrointestinal disorders) | 8 | 4
Constipation (Gastrointestinal disorders) | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Oral pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 6 | 3
Pyrexia (General disorders) | 3 | 2
Chills (General disorders) | 0 | 3
Asthenia (General disorders) | 1 | 0
Catheter site rash (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Injection site erythema (General disorders) | 1 | 0
Injection site rash (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 3
Dizziness (Nervous system disorders) | 3 | 3
Dysgeusia (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 0 | 2
Intercranial aneurysm (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 3
Platelet count decreased (Investigations) | 0 | 5
White blood cell count decreased (Investigations) | 0 | 4
Blood bilirubin increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Amylase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Protein total decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Rash pustular (Infections and infestations) | 1 | 2
Folliculitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Vulvitis (Infections and infestations) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Vision blurred (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 1 | 0
Corneal opacity (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT02706899/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT02706899/SAP_001.pdf